CLINICAL TRIAL: NCT05474937
Title: Nasal Inhalation of Sevoflurane Versus Midazolm,Ketamine and Propofol For Pediatric Undergoing Upper Gastrointestinal Endoscopy
Brief Title: Inhalation of Sevoflurane Versus Intravenous Midazolam,Ketamine,Propofol For Pediatrics Undergoing Upper GI Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Salih Salim Salih Bahri, Resident of anesthesia and intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9535
Record Dates: First submitted 2022-07-06; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Upper GI Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Midazolam; Ketamine; Propofol

STUDY DESIGN:
Intervention Model Description: prospective randomized clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inhalational Sevoflurane (Active Comparator): In the field of pediatric gastroenterology, upper gastrointestinal endoscopy has established itself as a diagnostic and therapeutic tool. In order to increase patient tolerance during this procedure, deep sedation is essential. Children are at a higher risk of serious adverse effects from procedural sedation; thus, their safety is a primary issue throughout this procedure. Multiple studies have been done to find the ideal method for procedural sedation in terms of ease of administration, quality, safety of sedation and recovery profile, but the consensus seems lacking. In this study we will compare between nasal inhalation of sevoflurane versus intravenous ketamine, midazolam and propofol for pediatrics undergoing upper gastrointestinal endoscopy.
  Interventions: Drug: Sevoflurane Inhalation Solution; Drug: Midazolam, Ketamine and Propofol
- Intravenous Ketamine, Midazolam and Propofol group (Active Comparator): Preoxygenation with 100% O2 for 1 minute, by proper sized face mask. Patients in Ketamine -midazolam -propofol (KMP) group will receive 1-1.5 mg/kg IV ketamine and 0.05mg/kg IV Midazolam and 1mg/kg IV Propofol as induction dose then followed by incremental doses of 0.5 mg/kg IV Propofol alone for maintenance and if procedure is prolonged propofol infusion at 100 μg/kg/min is given for maintenance of sedation. Induction dose will be considered as adequate if adequate jaw relaxation for endoscope insertion and Modified Ramsay Sedation Score (MRSS) ≥7 occurs with maintenance of spontaneous respiration. Induction time will be considered as time from beginning of IV agent to achievement of MRSS ≥7. After endoscope insertion, maintenance of oxygenation by nasal cannula at flow twice the minute ventilation of the patient.
  Interventions: Drug: Sevoflurane Inhalation Solution; Drug: Midazolam, Ketamine and Propofol

INTERVENTIONS:
Drug: Sevoflurane Inhalation Solution — Patients in inhalational group will receive Sevoflurane at 7% dial concentration in 100% O2 by an appropriately sized face mask until adequate sedation occurs as adequate jaw relaxation for the endoscope insertion and attainment of Modified Ramsay Sedation Score (MRSS) 7 (i.e., Asleep, reflex withdrawal to painful stimuli only).
Drug: Midazolam, Ketamine and Propofol — Preoxygenation with 100% O2 for 1 minute, by proper sized face mask. Patients in Ketamine -midazolam -propofol (KMP) group will receive 1-1.5 mg/kg IV ketamine and 0.05mg/kg IV Midazolam and 1mg/kg IV Propofol as induction dose then followed by incremental doses of 0.5 mg/kg IV Propofol alone for maintenance and if procedure is prolonged propofol infusion at 100 μg/kg/min is given for maintenance of sedation. Induction dose will be considered as adequate if adequate jaw relaxation for endoscope insertion and Modified Ramsay Sedation Score (MRSS) ≥7 occurs with maintenance of spontaneous respiration. Induction time will be considered as time from beginning of IV agent to achievement of MRSS ≥7. After endoscope insertion, maintenance of oxygenation by nasal cannula at flow twice the minute ventilation of the patient

SUMMARY:
In the field of pediatric gastroenterology, upper gastrointestinal endoscopy has established itself as a diagnostic and therapeutic tool. In order to increase patient tolerance during this procedure, deep sedation is essential. Children are at a higher risk of serious adverse effects from procedural sedation; thus, their safety is a primary issue throughout this procedure. Multiple studies have been done to find the ideal method for procedural sedation in terms of ease of administration, quality, safety of sedation and recovery profile, but the consensus seems lacking. In this study we will compare between nasal inhalation of sevoflurane versus intravenous ketamine, midazolam and propofol for pediatrics undergoing upper gastrointestinal endoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. A consent from the parents or 1st degree relative.
2. Both sexes.
3. Pediatric patients aged 1year to 4 years old undergoing
4. elective upper GI endoscopy.
5. ASA class I &II.
6. BMI between 5th percentile and the 85th percentile (http://www.kidshealth.org).

Exclusion Criteria:

1. Hypersensitivity to drugs included in the study.
2. Difficult airway or known airway problems.
3. Active bleeding from esophageal varices.
4. Respiratory and cardiac problems.
5. Neurological disorders

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
sedative effect | 1 hour
  Sedative effect will be assessed in terms of induction time success of induction and maintenance

SECONDARY OUTCOMES:
adverse events | 2 hours
  Safety will be assessed in terms of occurrence of complications

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication
Access Criteria: contact the principle investigator

REFERENCES:
- [Background] Agostoni M, Fanti L, Gemma M, Pasculli N, Beretta L, Testoni PA. Adverse events during monitored anesthesia care for GI endoscopy: an 8-year experience. Gastrointest Endosc. 2011 Aug;74(2):266-75. doi: 10.1016/j.gie.2011.04.028. Epub 2011 Jun 25. PMID 21704990
- [Background] Agrawal D, Feldman HA, Krauss B, Waltzman ML. Bispectral index monitoring quantifies depth of sedation during emergency department procedural sedation and analgesia in children. Ann Emerg Med. 2004 Feb;43(2):247-55. doi: 10.1016/s0196-0644(03)00721-2. PMID 14747816
- [Background] Basturk A, Artan R, Yilmaz A. Efficacy and safety of midazolam and ketamine in paediatric upper endoscopy. Arab J Gastroenterol. 2017 Jun;18(2):80-82. doi: 10.1016/j.ajg.2017.05.004. Epub 2017 Jun 1. PMID 28579345
- [Background] Biliskov AN, Ivancev B, Pogorelic Z. Effects on Recovery of Pediatric Patients Undergoing Total Intravenous Anesthesia with Propofol versus Ketofol for Short-Lasting Laparoscopic Procedures. Children (Basel). 2021 Jul 19;8(7):610. doi: 10.3390/children8070610. PMID 34356589
- [Background] Gaya da Costa M, Kalmar AF, Struys MMRF. Inhaled Anesthetics: Environmental Role, Occupational Risk, and Clinical Use. J Clin Med. 2021 Mar 22;10(6):1306. doi: 10.3390/jcm10061306. PMID 33810063
- [Background] Oh C, Kim Y, Eom H, Youn S, Lee S, Ko YB, Yoo HJ, Chung W, Lim C, Hong B. Procedural Sedation Using a Propofol-Ketamine Combination (Ketofol) vs. Propofol Alone in the Loop Electrosurgical Excision Procedure (LEEP): A Randomized Controlled Trial. J Clin Med. 2019 Jun 28;8(7):943. doi: 10.3390/jcm8070943. PMID 31261820